CLINICAL TRIAL: NCT06546540
Title: Evaluator Blind, Controlled, Preliminary Clinical Study of Telitacicept in the Treatment of Diffuse Systemic Sclerosis With Progressive Skin Progression
Brief Title: The Safety and Efficacy of Telitacicept in the Treatment of Systemic Sclerosis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Mu Rong, professor, Peking University Third Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BYSYDL2021005
Record Dates: First submitted 2024-08-04; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — telitacicept

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telitacicept (Experimental)
  Interventions: Drug: Telitacicept
- Conventional (No Intervention)

INTERVENTIONS:
Drug: Telitacicept — 160mg，once weekly
  Arms: Telitacicept

SUMMARY:
Systemic sclerosis (SSc) is a chronic, multisystem autoimmune disease characterized by potentially widespread and progressive skin fibrosis and vascular abnormalities, and may involve the musculoskeletal, gastrointestinal, pulmonary, cardiac, renal, neuromuscular, and urogenital systems. At present, there is no clear and effective drug treatment for the progression of scleroderma skin lesions, and there is a lack of authoritative treatment recommendations. In recent years, research on the treatment of B cells in SSc suggests that targeted B cell therapy has certain safety and effectiveness for SSc patients. Telitacicept is a fully human fusion protein that is a fusion of TACI protein and IgG1 protein. Telitacicept can inhibit the further development and maturation of immature B cells by blocking BLyS. At the same time, Telitacicept can also inhibit the differentiation of mature B cells into plasma cells by blocking APRIL, and affect the secretion of abnormal self reactive plasma cell autoantibodies, better controlling disease activity. The effectiveness and safety of SSc treatment require further research. This study is an evaluator blind, parallel controlled clinical trial that included 20 SSc patients who still had skin progression despite conventional treatment. The patients were divided into two groups, one group included patients who did not improve with conventional treatment for skin lesions, and the other group included patients who received traditional conventional treatment. The main outcome of the study was to evaluate the efficacy and safety of Telitacicept in the treatment of progressive skin lesions in SSc, and the secondary outcome was to evaluate the impact of Telitacicept on lung function, gastrointestinal symptoms, pulmonary arterial hypertension, disease activity, and quality of life in SSc.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with systemic sclerosis who met the ACR2013 classification criteria for systemic sclerosis and approved this trial
2. Age: 18 years or older
3. Lung function FVC% > 50%
4. Positive for ANA or scleroderma related autoantibodies
5. Patients with disease activity after conventional treatment: new skin involvement or deterioration of two new body areas or skin thickening and deterioration after 6 months of conventional treatment (δMRSS ≥0 points)
6. The dose of the following drugs was stable for at least 6 months before the first use of the study drug: mycophenolate mofetil, cyclophosphamide；First use of study drug precorticosteroids (≤10 mg prednisone/day or equivalent) for at least 30 days

Exclusion Criteria:

1. Subjects who did not consent to participate in the clinical trial
2. Subjects with mixed connective tissue disease or overlap syndrome
3. Focal scleroderma
4. Pregnant women, lactating women and men or women who have planned to have children in the last 12 month
5. Allergic reaction: History of allergy to human derived biological products
6. Participants who had participated in any clinical trial within 28 days prior to initial screening/or within a 5-fold half-life of the study compound (whichever is longer)
7. Those who have received live vaccine in the last month
8. B cell-targeted therapies such as rituximab, iparizumab, and beliumab were used within one year
9. Tumor necrosis factor inhibitors and interleukin-receptor blockers were used within one year.
10. Patients who used intravenous gamma globulin (IVIG), prednisone ≧100 mg/d for more than 14 days within one month or underwent plasma exchange surgery
11. Use Chinese medicine for treatment within one month
12. There is active infection (such as herpes zoster, HIV infection, active tuberculosis, etc.) during the screening period
13. There are serious complications such as uncontrolled congestive heart failure, arrhythmias, severe pulmonary hypertension or hypertension, severe gastrointestinal involvement, liver function impairment, active infection, severe diabetes mellitus, atherosclerotic heart disease, malignancy, AIDS, or severe peripheral vascular disease.
14. Patients with severe depression, psychosis or suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-08 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Changes of mRSS in patients after 52 weeks of treatment | base line and week 52
  The range and degree of skin thickening can be evaluated using the modified Rodnan skin score (mRSS) . The evaluator palpated 17 areas of the patient's body, and calculated the skin thickness of each area on a scale of 0-3 points, with a total score of 51 points. The skin progression was evaluated through changes in mRSS scores.
The safety of Telitacicept | up to 52 weeks
  Evaluate adverse drug reactions

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No